CLINICAL TRIAL: NCT06525324
Title: Comparing The Effectiveness Of T-PRF And PRF With Bone-Graft[DMBM]TM Around Immediate Implants - A RANDOMISED CONTROL TRIAL
Brief Title: Comparision of Clinical Efficacy of Immediate Implants With T-PRF and Bone-graft Versus PRF and Bone-graft
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02_D012_00041
Record Dates: First submitted 2024-07-19; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Dental Implants
Keywords: PRF with bone graft; T-PRF with bone graft
MeSH Terms: interventions — Transplantation, Heterologous; Prolactin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- in 10 sites immediate implant will be placed along with T-PRF and xenograft (Experimental): Immediate implant is placed along with T-PRF and xenograft.
  Interventions: Procedure: Immediate implant surgery with T-PRF and xenograft
- in 10 sites immediate implants will be placed with PRF and xenograft (Active Comparator): Immediate implant is placed along with PRF and xenograft as control
  Interventions: Procedure: Immediate implant surgery with PRF and xenograft

INTERVENTIONS:
Procedure: Immediate implant surgery with T-PRF and xenograft — A mucoperiosteal flap will be raised and atraumatic extraction will be done. An immediate implant with T-PRF and xenograft will be placed according to the standard protocol.
  The surgical wound closure will be coapted with mattress and single interrupted sutures
  Arms: in 10 sites immediate implant will be placed along with T-PRF and xenograft
Procedure: Immediate implant surgery with PRF and xenograft — A mucoperiosteal flap will be raised and atraumatic extraction will be done. An immediate implant with PRF and xenograft will be placed according to the standard protocol .
  The surgical wound closure will be coapted with mattress and single interrupted sutures
  Arms: in 10 sites immediate implants will be placed with PRF and xenograft

SUMMARY:
The normal architecture of the alveolar process is altered by periodontitis, which also causes the loss of alveolar bone surrounding the teeth. Untreated periodontitis may cause teeth to become mobile and leads to loss of teeth.

In such cases, one of the treatment modalities is extraction of the tooth and placement of immediate implant which reduces the waiting period. And due to the resorption of alveolar ridge the bone graft will be used along with T-PRF and PRF.

So this study aims at the placement of immediate implants along with T-PRF with bone graft and PRF with bone graft.

DETAILED DESCRIPTION:
Dental implants have become more common treatment for replacing missing teeth and aim to improve chewing efficiency, physical health and esthetic. And their will be resorption of alveolar process due to periodontitis . In such compromised cases, to achieve bone augmentation around immediately placed implants a new modality of using platelet rich fibrin (PRF) along with graft material has gained considerable interest.

Successful clinical results have been reported with L-PRF, but some physicians worry about a possible health hazard with glass-evacuated blood collection tubes with silica activators. O'Connell described the unavoidable silica contact. The silica particles in the tube, although dense enough to sediment with the red blood cells, are small enough for a fraction to remain colloidally suspended in the buffy coat, fibrin, and platelet-poor plasma layers therefore, these particles might reach the patient when the product is used for treatment.

Recently use of titanium tubes in the preparation of PRF showed more polymerized fibrin formation with longer resorption in tissues as titanium seems to be more effective in activating platelets than silica and also eliminates the possible silica contamination.

The use of T-PRF(Titanium PRF) along with xenograft creates a block graft with high concentrated growth factors, platelets and leucocytes which enhance development of bone and eliminates the possible silica contamination.

Hence, the aim of the study is to compare the effectiveness of T-PRF with xenograft [DMBM] and PRF with xenograft [DMBM] around immediate implants.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18-55 years of age.
2. Presence of non-restorable teeth (maxillary or mandibular) due to trauma, decayed, mobility, root resorption, root stumps, root fracture, over retained deciduous tooth, endodontic or periodontal failure in whom immediate implants can be placed.
3. Good oral hygiene.
4. Good patient compliance.
5. Class I extraction socket defects according to modified Elian et al 2021.

Exclusion Criteria:

1. Systemic complications (uncontrolled diabetes and severe cardiovascular or infectious diseases).
2. Intravenous and oral bisphosphonate therapy.
3. Patients who are psychologically unable to participate.
4. Pregnant and lactating participants with bone diseases
5. Patients on chemotherapy or radiotherapy
6. Alcohol or drug abuse.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Marginal Bone Level Using RVG and Grid. | Baseline , 3 months , 9 months
  Marginal bone level measured .
Soft tissue healing | Baseline ,3 months , 9 months
  Soft tissue healing will be assessed using Wachtel-et-al 2009 classification
Bone fill using RVG with grid | 3 months , 9 months
  Measuring the Bone fill by formula Linear bone growth/depth of original bone defect
Bone dimensions using CBCT | 9 months
  Extent of bone dimensions is measured through CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Krishnadevaraya college of dental sciences, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared with other researchers.

REFERENCES:
- [Background] Tunali M, Ozdemir H, Kucukodaci Z, Akman S, Firatli E. In vivo evaluation of titanium-prepared platelet-rich fibrin (T-PRF): a new platelet concentrate. Br J Oral Maxillofac Surg. 2013 Jul;51(5):438-43. doi: 10.1016/j.bjoms.2012.08.003. Epub 2012 Aug 28. PMID 22951383